CLINICAL TRIAL: NCT03752164
Title: Kids 2 Be & Breathe: A Study on the Use of Yoga and Mindfulness in Children With Severe Asthma
Brief Title: Kids 2 Be & Breathe: A Study on the Use of Yoga and Mindfulness in Children With Severe Asthma (K2B2)
Acronym: K2B2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM20014054
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga and Mindfulness (Experimental): An intervention consisting of one session lasting 30 minutes where a certified yoga instructor teaches the children gentle yoga and mindfulness skills.
  Interventions: Behavioral: Yoga and Mindfulness Skills

INTERVENTIONS:
Behavioral: Yoga and Mindfulness Skills — Single brief session in which children are taught yoga and skills in mindfulness

SUMMARY:
This proposed pilot study will examine the tolerability, feasibility, acceptability, and preliminary effects of a gentle yoga intervention "Kids 2 Be & Breathe" (K2B2; a manualized 30 minute gentle yoga and mindfulness session held one-on-one) in urban children aged 7-11 with severe asthma.

DETAILED DESCRIPTION:
Pre-Intervention Assessment: permission/assent from the child and consent of the parent/guardian will be obtained and initial data and measurements will be collected to ensure continued eligibility; baseline measures will be assessed.

Intervention: participants will engage in a one-time manualized, age appropriate, 1:1, 30-minute intervention involving gentle yoga and mindfulness techniques in a private room in the Pediatric Research Unit at the Children's Hospital of Richmond. The intervention will be taught by certified and experienced child yoga instructors who have been trained in the study protocol by the applicant. These yoga instructors collaborated with the interdisciplinary research team in the development of manualized age-appropriate yoga sequences. Parents/guardians will be invited to observe the yoga session. Intervention fidelity will be maintained through the use of a manualized intervention and the PI observing all sessions for manual consistency. The intervention will cease if the participant suffers from any asthma symptoms during the intervention, such as wheezing, coughing, retractions, accessory muscle use, chest tightness or shortness of breath, or experiences any other adverse events which precludes the his or her ability to actively participate in the intervention.

Post-Intervention Assessment: upon completion of the intervention, brief semi-structured interviews will be conducted with the child and parent/guardian separately in order to explore the acceptability of the intervention and the PI will again assess the child for any asthma symptoms or adverse events. Post-intervention pulmonary function test and vital sign measurements will then be collected.

ELIGIBILITY:
Inclusion Criteria:

* on medium to high doses of steroids and/or leukotriene inhibitors
* a Child-Asthma Control Test Score <21

Exclusion Criteria:

* inability to speak English (child); inability to read/write English (parent/guardian)
* child hospitalized in past two weeks for their asthma
* current illness associated with oral temperature >100.4
* pulse ox <95% and/or any wheezing, retractions or accessory muscle use

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Tolerability: FEV1%(forced expiratory volume in 1 second ) asthma symptoms and adverse events | 2 hours
  whether intervention causes an exercise induced bronchoconstriction, asthma symptoms or adverse events

SECONDARY OUTCOMES:
Preliminary Effects: Change in FEV1 | Baseline to 2 hours
  measuring the change in FEV1 pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Lack, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No